CLINICAL TRIAL: NCT02912429
Title: Onlay- vs. Inlay-Type Patellofemoral Arthroplasty: a Prospective, Comparative Study
Brief Title: Onlay vs. Inlay Patellofemoral Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Michael Liebensteiner, Principal Investigator and Coordinating Investigator, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PF-Arthroplasty 1
Record Dates: First submitted 2016-09-13; First posted 2016-09-23 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Patellofemoral Joint; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Inlay (Other): specific technical type of patellofemoral arthroplasty
  Interventions: Device: Patellofemoral Arthroplasty
- Onlay (Other): specific technical type of patellofemoral arthroplasty
  Interventions: Device: Patellofemoral Arthroplasty

INTERVENTIONS:
Device: Patellofemoral Arthroplasty

SUMMARY:
There is currently no sufficient evidence if there is superiority of one of the two available types (onlay type, inlay type) of patellofemoral arthroplasty. Therefore, it is the aim of this study to compare the two types in a prospective comparative setting. Patients on the waiting list for patellofemoral arthroplasty are randomized to either onlay or inlay type patellofemoral arthroplasty. The KOOS - knee score serves as the primary outcome parameter. Secondary outcome parameters are the Marx Activity Scale, the HSS patella score, the Kujala Score, radiographic loosening, progression of tibiofemoral degeneration, revision surgery and parameters of patellofemoral tracking. Inferential statistics will be performed at 1-year follow up data-sets.

ELIGIBILITY:
Inclusion Criteria:

* patellofemoral osteoarthritis, waiting list for patellofemoral arthroplasty

Exclusion Criteria:

* systemic inflammatory arthropathy
* tibiofemoral joint degeneration IKDC grade C or worse
* severe degeneration of also the trochlea margins (inlay PFA not adequate)
* patellectomy
* previous implantation of tibiofemoral metal implants
* extension loss >5 degree
* knee flexion of less than 100°
* planned concomitant tibiofemoral procedures (eg. coronal plane osteotomies, tibiofemoral cartilage procedures, tibiofemoral ligament procedures)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
KOOS knee score | 1 year

SECONDARY OUTCOMES:
Kujala Score | 1 year
Marx Activity Scale | 1 year
HSS patella Score | 1 year

OTHER OUTCOMES:
radiolucent lines adjacent to the prosthesis | 20 years
  radiolucent lines adjacent to the prosthesis indicate prosthesis loosening
revision of prosthesis | 20 years
  reoperations with ex/implantation of implants are defined as prosthetic revision
progression of tibiofemoral osteoarthritis | 20 years
  progression of tibiofemoral osteoarthritis is assessed in terms of IKDC grades A-D

CONTACTS AND LOCATIONS:
Overall Officials: michael liebensteiner, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria